CLINICAL TRIAL: NCT06120296
Title: Effect of the Hypotension Prediction Index on the Prevalence of Intra-operative Hypotension During Shoulder Surgery in Beach Chair: A Prospective Randomized Clinical Trial.
Brief Title: Hypotension Prediction Index for Shoulder Surgery in Beach Chair.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Geertrui Dewinter (Other)
Responsible Party: Sponsor-Investigator, Geertrui Dewinter, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: GDW 10/2022
Record Dates: First submitted 2023-10-12; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hypotension During Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): In the blinded HPI group (the control group) the arterial waveform and pressure will be presented on a Philips patient monitor (the standard monitor), while the display of the hemosphere monitor shall be covered and the alarms will be silenced.
- intervention group (Experimental): In the unblinded HPI group (the intervention group), the arterial waveform and pressure will be displayed on the anesthesia monitor and the HPI on the Hemosphere monitor of Edwards Lifesciences (the study monitor).
  Interventions: Device: Acumen Hypotension prediction Index software

INTERVENTIONS:
Device: Acumen Hypotension prediction Index software — In the unblinded HPI group (the intervention group), the arterial waveform and pressure will be displayed on the anesthesia monitor and the HPI on the Hemosphere monitor of Edwards Lifesciences (the study monitor).
  Arms: intervention group

SUMMARY:
The beach chair position is the most commonly used position during shoulder surgery and offers the surgeon numerous advantages over the lateral decubitus position. However, the beach chair position can also lead to hemodynamic changes, including hypotension and cerebral hypoperfusion. It is therefore the anesthesiologist's job to prevent hypotension during the procedure.

The Acumen Hypotension Predictor Index or HPI for short is a software program that can predict the occurrence of low blood pressure during surgery shortly before it occurs. Studies have already demonstrated the effectiveness of HPI in various operations, where hypotension is defined as a mean arterial blood pressure < 65mmHg for at least 1 minute. To our knowledge, the low blood pressure prediction index has not yet been investigated for the prevention of low blood pressure in shoulder surgery in the beach chair position.

The HPI is built into a monitor that is switched on in addition to the standard monitoring for monitoring blood pressure, pulse, saturation, among other things. The monitor gives a signal when an episode of low blood pressure will occur within 15 minutes. This gives the anesthesiologist the opportunity to anticipate in time so that the occurrence of low blood pressure can be avoided.

Goal The aim of this study is to evaluate the efficacy of the HPI in predicting and reducing the incidence of hypotension during shoulder surgery in the beach chair position.

Procedure A total of 144 patients will participate in this study. Patients will be randomized to the intervention group or the control group according to a 1:1 allocation. In addition to standard monitoring, the HPI monitor will be turned on for all patients. For patients in the control group, the HPI monitor screen will be blinded and the alarms muted.

Patients between 18 and 85 years of age with a BMI ≤ 40 kg/m2 undergoing elective shoulder surgery are eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 40 kg/m2
* Patient can give informed consent
* ASA I-IV
* Invasive blood monitoring
* General anesthesia combined with interscalene block

Exclusion Criteria:

* - Refusal of participation
* Hypotension before surgery (MAP< 65 mmHg)
* History of stroke
* Dementia
* Contra-indication for interscalene block
* Contra-indication for general anesthesia
* Dialysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Time-weighted average MAP< than 65 mmHg | during surgery
  Calculated as depth of hypotension below a MAP of 65 mmHg x time spent below a MAP of 65 mmHg (in minutes) divided by total duration of anesthesia (in minutes))

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesie Research, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No